CLINICAL TRIAL: NCT03883906
Title: Donor-Derived Viral Specific T-cells (VSTs) for Prophylaxis Against Viral Infections After Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoxworth Blood Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0229
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Allogeneic Stem Cell Transplant; Viral Infection
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viral Specific T-cells (VSTs) (Experimental)
  Interventions: Biological: Viral Specific T-cells (VSTs)

INTERVENTIONS:
Biological: Viral Specific T-cells (VSTs) — VSTs will be infused into stem cell transplant recipients

SUMMARY:
The purpose of this research study is to learn more about the use of viral specific T-lymphocytes (VSTs) to prevent viral infections that may happen after allogeneic stem cell transplant. Allogeneic means the stem cells come from another person. VSTs are cells specially designed to fight viral infections that may happen after a stem cell transplant (SCT).

Stem cell transplant reduces your ability to fight infections. Viral infections are a common problem after transplant and can cause significant complications. Moreover, treatment of viral infections is expensive and time consuming, with families often administering prolonged treatments with intravenous anti-viral medications, or patients requiring prolonged admissions to the hospital. The medicines can also have side effects like damage to the kidneys or reduction in the blood counts, so in this study we are trying to find a way to prevent these infections.

ELIGIBILITY:
Inclusion Criteria:

* Recipient must be at least 21 days after stem cell infusion
* Clinical status must allow tapering of steroids to < 0.5mg/kg prednisone or other steroid equivalent

Exclusion Criteria:

* Patients who have developed viral infection or reactivation will be ineligible for prophylactic infusions of VSTs
* Active acute GVHD grades II-IV
* Uncontrolled relapse of malignancy
* Infusion of ATG or alemtuzumab within 2 weeks of VST infusion. Additionally, in patients who received alemtuzumab as part of their conditioning regimen, alemtuzumab levels will be collected in the second week following stem cell infusion. The level must be less than, or equal to, 0.15 prior to infusion of VSTs. In patients with level greater than 0.15, alemtuzumab levels can be checked serially until a level ≤ 0.15 is obtained. They would become eligible for prophylactic VST infusion at that point if there is still no evidence of viral infection at that time.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grimley, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Viral Specific T-cells (VSTs)
Started | 30
Completed | 23
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Viral Specific T-cells (VSTs)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of a Toxicity
Description: Participants will be assessed for the presence of a toxicity.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Specific T-cells (VSTs)
Number analyzed (Participants) | 23
Participants | 0

2. Primary Outcome: Number of Participants With Acute Graft-Vs-Host Disease (aGVHD)
Description: Participants will be assessed for the presence of aGVHD.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Specific T-cells (VSTs)
Number analyzed (Participants) | 23
Participants | 2

3. Secondary Outcome: Number of Participants With Presence of a Viral Infection
Description: Participants will be assessed for the presence of viral infection.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Specific T-cells (VSTs)
Number analyzed (Participants) | 23
Participants | 14

ADVERSE EVENTS:
Time Frame: 30 days
Description: All adverse events that occur from the administration of first VST infusion through 30 days after the last VST infusion were recorded per the protocol. Events occurring greater than 30 days after the last VST infusion were assessed and recorded only when they are unexpected and determined to be at least possibly related to the VST infusion through 1 year after the last VST infusion.
Arm/Group | Viral Specific T-cells (VSTs)
All-Cause Mortality (participants affected / at risk) | 2/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viral Specific T-cells (VSTs) (N=23)
GVHD, skin (Skin and subcutaneous tissue disorders) | 1 (1)
GVHD, stomach (Gastrointestinal disorders) | 1 (1)
GVHD, sigmoid colon & rectum (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT03883906/Prot_001.pdf